CLINICAL TRIAL: NCT03057756
Title: Nine Months' Short Course Regimen Protocol for the Treatment of Multidrug Resistance-tuberculosis (MDR-TB) Patients in Gabon
Brief Title: Treatment of Tuberculosis Multidrug Resistance Treatment of Tuberculosis Multidrug Resistance
Acronym: TB-MR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Collaborators: Institute of Tropical Medicine, University of Tuebingen (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Ayola Akim ADEGNIKA, Professor, Centre de Recherche Médicale de Lambaréné
Other Study IDs: TB-MR 001/2015
Record Dates: First submitted 2017-02-13; First posted 2017-02-20 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Multi-drug Resistant Tuberculosis
Keywords: Multi-drug Resistant Tuberculosis; short course regimen protocol
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — Protons

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TB-MR patients: Patients older than 15 years old receiving Km+ Mfx+ Pto + H + Cfz +E+Z
  Interventions: Combination Product: Km+ Mfx+ Pto + H + Cfz +E+Z

INTERVENTIONS:
Combination Product: Km+ Mfx+ Pto + H + Cfz +E+Z — Second generation of anti tuberculosis Kanamycine, Moxifloxacine,Prothionamide, isoniazide,Clofazimine, Ethambutol,Pyrazinamide

SUMMARY:
The principal objective is to evaluate a cure rate and number of adverse events of with confirmed multidrug-resistant tuberculosis patient treated with a 9months regimen.

DETAILED DESCRIPTION:
Study participants will be followed up, under existing protocol derived from a study protocol developed by the "Union internationale contre les maladies respiratoires" and carried out already in 9 Africans countries. Participants will be hospitalised for at least four month, period which they will be given treatments, assessed for adverse events, monitored for TB-MR strains using culture techniques, at the monthly basis. If patients found with negative sputum culture at month four they will be dischrged from the hospital, and then treated four an additional five montns and then follow up, clinically and biologically for an additional six months before being declared as cured.

ELIGIBILITY:
Inclusion criteria:

* Aged 15 years and above
* Never been treated with second line anti-TB drugs for more than one month,
* Give written consent to participate
* Agree to be hospitalised for at least four months in specialised healthcare
* Willing to adhere to ambulatory directly observed treatment by a healthcare worker;

Exclusion criteria:

* Pregnant during inclusion process
* Presented with altered clinical status condition as judged by the clinician
* Knowing of history of hypersensitivity reaction to any of the drugs to be used
* Baseline ECG does not show a QT space superior to 500ms
* Refusal to participate into study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: study population will consist of all consecutive patients with bacteriologically proven MDR-TB who fulfil the inclusion criteria .
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2015-09-11 (Actual); Primary Completion 2023-04-04 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
cure rate post treatment | Six months post treatment
  Proportion of participants alive and presented with negative sputum culture for TB and with the absence of clinical, X-Ray and biological disorders related to TB

SECONDARY OUTCOMES:
TB-culture | 4 months after start of the treatment
  First TB culture negative time
Regimen tolorability | Throughout treatment period (9months)
  treatment, safety through clinical and biological assessment
Adverse events | duration of participant in the study (15months)
  solicited and unsolicited adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ayola A Adegnika, MD, PhD, Principal Investigator — Centre de Recherches Médicales de Lambaréné
Locations (1):
- Centre de Recherches Médicales de Lambaréné, Lambaréné, Please Select, Gabon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eurosurveillance editorial team. WHO revised definitions and reporting framework for tuberculosis. Euro Surveill. 2013 Apr 18;18(16):20455. No abstract available. PMID 23611033
- [Result] Pablos-Mendez A, Raviglione MC, Laszlo A, Binkin N, Rieder HL, Bustreo F, Cohn DL, Lambregts-van Weezenbeek CS, Kim SJ, Chaulet P, Nunn P. Global surveillance for antituberculosis-drug resistance, 1994-1997. World Health Organization-International Union against Tuberculosis and Lung Disease Working Group on Anti-Tuberculosis Drug Resistance Surveillance. N Engl J Med. 1998 Jun 4;338(23):1641-9. doi: 10.1056/NEJM199806043382301. PMID 9614254
- [Result] Falzon D, Jaramillo E, Schunemann HJ, Arentz M, Bauer M, Bayona J, Blanc L, Caminero JA, Daley CL, Duncombe C, Fitzpatrick C, Gebhard A, Getahun H, Henkens M, Holtz TH, Keravec J, Keshavjee S, Khan AJ, Kulier R, Leimane V, Lienhardt C, Lu C, Mariandyshev A, Migliori GB, Mirzayev F, Mitnick CD, Nunn P, Nwagboniwe G, Oxlade O, Palmero D, Pavlinac P, Quelapio MI, Raviglione MC, Rich ML, Royce S, Rusch-Gerdes S, Salakaia A, Sarin R, Sculier D, Varaine F, Vitoria M, Walson JL, Wares F, Weyer K, White RA, Zignol M. WHO guidelines for the programmatic management of drug-resistant tuberculosis: 2011 update. Eur Respir J. 2011 Sep;38(3):516-28. doi: 10.1183/09031936.00073611. Epub 2011 Aug 4. PMID 21828024
- [Result] Stolp SM, Huson MA, Janssen S, Beyeme JO, Grobusch MP. Tuberculosis patients hospitalized in the Albert Schweitzer Hospital, Lambarene, Gabon-a retrospective observational study. Clin Microbiol Infect. 2013 Nov;19(11):E499-501. doi: 10.1111/1469-0691.12278. Epub 2013 Jul 4. PMID 23826878
- [Result] Van Deun A, Maug AK, Salim MA, Das PK, Sarker MR, Daru P, Rieder HL. Short, highly effective, and inexpensive standardized treatment of multidrug-resistant tuberculosis. Am J Respir Crit Care Med. 2010 Sep 1;182(5):684-92. doi: 10.1164/rccm.201001-0077OC. Epub 2010 May 4. PMID 20442432
- [Result] Laserson KF, Thorpe LE, Leimane V, Weyer K, Mitnick CD, Riekstina V, Zarovska E, Rich ML, Fraser HS, Alarcon E, Cegielski JP, Grzemska M, Gupta R, Espinal M. Speaking the same language: treatment outcome definitions for multidrug-resistant tuberculosis. Int J Tuberc Lung Dis. 2005 Jun;9(6):640-5. PMID 15971391
- [Result] Chiang CY, Caminero JA, Enarson DA. Reporting on multidrug-resistant tuberculosis: a proposed definition for the treatment outcome 'failed'. Int J Tuberc Lung Dis. 2009 May;13(5):548-50. No abstract available. PMID 19383184
- [Result] World Health Organization; International Union Against Tuberculosis and Lung Disease; Royal Netherlands Tuberculosis Association. Revised international definitions in tuberculosis control. Int J Tuberc Lung Dis. 2001 Mar;5(3):213-5. No abstract available. PMID 11326818
- See also: web based information — http://apps.who.int//iris/handle/10665/66368